CLINICAL TRIAL: NCT04380844
Title: Effects of an Activity Control System in Patients With Diabetes: a Randomized
Brief Title: Effects of an Activity Control System in Patients With Diabetes: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: orcid.org/0000-0002-869
Record Dates: First submitted 2020-04-04; First posted 2020-05-08 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: artificial intelligence; diabetes mellitus; self-care; telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beprevent (Active Comparator): 10 will become part of the intervention group. Each of the participants in the intervention group is selected. At first, they are given a series of questionnaires, later (1 day later) we stay at their home to install the Beprevent device, which will remain in their home for a period of two weeks, to finish and once the device of your home, we will proceed to pass the same questionnaires as at the beginning of the test, in order to compare results.
  Interventions: Other: Beprevent
- patients only evaluated (No Intervention): 10 will be included in the control group. During the period of the study, we will pass the same questionnaires in the participants assigned to the control group, also leaving a time interval of two weeks, and no device will be installed, nor will any monitoring be carried out in their homes.

INTERVENTIONS:
Other: Beprevent — 10 will become part of the intervention group. At first, they are given a series of questionnaires, later (1 day later) we stay at their home to install the Beprevent device, which will remain in their home for a period of two weeks, to finish and once the device of your home, we will proceed to pass the same questionnaires as at the beginning of the test, in order to compare results.
  Arms: Beprevent

SUMMARY:
Using a smart device (Beprevent) to monitor activities of daily living improves the lifestyle of patients with DM2

DETAILED DESCRIPTION:
A 6-month randomized clinical trial to evaluate a home activity control system (Beprevent) in the management of the patient with DM2, through the individualized labeling of objects related to them. The study will include 20 patients with DM2 (10 in the intervention group and 10 in the control group) who live alone or with people who can´t move on their own. Data will be recorded to measure the degree of satisfaction of professionals and participants in the study, and clinical and epidemiological data at the start of the study (in its baseline situation) and at the end of the study (at 6 months), to assess the changes produced and Compare them between both study groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years, with the ability to give informed consent
* Patient who has autonomy to carry out activities of daily living (Barthel = 100)
* patient diagnosed with Diabetes Mellitus
* patient in pharmacological treatment
* To live alone or with a person who cannot move on their own
* they do not plan to change their address in the 6 months after inclusion in the study

Exclusion Criteria:

• DM2 patients whose most recent HbA1c value is ≤7%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Knowledge Questionnaire | 15 minuts
  The Diabetes Knowledge Questionnaire (DKQ-24) is a questionnaire made up of 24 questions about basic knowledge of the disease (10 items), glycemic control (7 items) and prevention of complications (7 items). The questions are closed, with answer options "yes, no and I don't know". Its maximum score is 24. The patient has better knowledge about diabetes the higher the score.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Gómez Lama, MD, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba; David Pérez Cruzado, Principal Investigator — Universidad Católica San Antonio de Murcia

IPD SHARING:
Plan to Share IPD: No